CLINICAL TRIAL: NCT04769492
Title: #ChopViolence/#ChopHIV: A Tailored Violence Prevention Intervention for Black Young MSM and Transgender Women From the House Ball Community to Improve HIV Outcomes and Decrease Exposure to Violence
Brief Title: #ChopViolence/#ChopHIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hektoen Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5R34MH121968 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-24 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Violence; HIV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Intervention (Other): Tailored violence prevention intervention (#ChopViolence/#ChopHIV) for B-YGBMSM and B-TW in the Chicago HBC.
  Interventions: Other: #ChopViolence/#ChopHIV

INTERVENTIONS:
Other: #ChopViolence/#ChopHIV — Tailored, community-based violence prevention intervention

SUMMARY:
Black young gay, bisexual and other men who have sex with men (B-YGBMSM) and transgender women (B-YTW) are disproportionately affected by HIV/AIDS in the U.S. Youth in the House Ball Community (HBC), a subculture of the Black gay community that offers a social network to freely express diverse sexual and gender identities, are among the most at-risk for HIV infection and loss to care, but barriers exist to the provision of HIV services within this community. One barrier is the increasing rates of violence. Interventions are needed that will interrupt the cycle of violence within the HBC to allow for adequate provision of HIV services and increased access to HIV care. The investigators propose to tailor the Cure Violence model for violence prevention for developmental-appropriateness, cultural-specificity and HIV relevance, then pilot test the new intervention (#ChopViolence/#ChopHIV) with B-YGBMSM and B-TW in the Chicago HBC. The proposed research activities will take place in six steps. In Step 1, the investigators will hold Youth Advisory Board meetings, finalize our assessment battery and conduct multiple baseline assessments (months 3, 9 & 15; n=75 per assessment point) at HBC venues to track trends in violence (i.e., intimate partner, HBC and neighborhood violence), HIV stigma, substance use, mental health, sexual risk and HIV care engagement. In Step 2, the investigators will employ ADAPT-ITT strategies for adapting evidence-based interventions including conducting a series of focus groups (n=32) with youth and leaders from the HBC in order to identify persuasive messaging around decreasing violence and improving HIV outcomes. Based on the focus group data as well as consultation with community experts, the investigators will then tailor the intervention to be relevant for the Chicago HBC and develop training materials along with standard operating procedures. In Step 3, the investigators will identify, recruit and train trusted members of the HBC to work as Violence Interrupters (VI) or Outreach Workers (OW). VI and OW will undergo training over the course of several weeks. Training activities include didactic seminars, webinars from the Cure Violence team, HIV education, conflict mediation skills and mock interruption and outreach activities. In Step 4, the investigators will pilot test the tailored intervention. VI will monitor HBC events as well as social media venues for potential violence and intervene. OW will build their client caseload with HIV+ youth identified as of highest-risk for violence and schedule sessions, phone calls, and assist with HIV care linkage. In Step 5, the investigators will conduct follow-up assessments (months 21, 27 & 33; n=75 per assessment point) at HBC events to continue to monitor trends in violence, HIV stigma, substance use, mental health, sexual risk and HIV care engagement. Qualitative interviews will be conducted with VI, OW and HIV+ intervention clients to explore the processes and strategies of intervention implementation, with a focus on implementation barriers and facilitators. Finally, in Step 6, the investigators will conduct data analysis, disseminate findings and produce scientific publications.

ELIGIBILITY:
Inclusion Criteria:

1. self-identified as Black,
2. ages 15-29
3. in attendance at a HBC event at the time of the assessment.

Exclusion Criteria:

-

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — cis-gender male or transgender female
Enrollment: 525 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Trauma History Questionnaire | last 12 months
  The Trauma History Questionnaire measures history of exposure to potentially traumatic events with 18 yes/no items addressing the occurrence of traumatic events in three categories: crime, general trauma, and sexual and physical assault experiences. We will adapt this measure for participants to identify if event occurred within HBC or within neighborhood.
Intimate Partner Violence | 12 months
  Intimate partner violence will be measured using a questionnaire developed for a multi-national study that consists of 4 questions that assess physical, emotional and sexual harm experienced by the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Cook County Health, Chicago, Illinois, United States